CLINICAL TRIAL: NCT06710847
Title: A Phase 1/2 First-Time-in-Human, Open-label, Multicenter, Dose Escalation and Expansion Study of the Oral DNA Helicase Werner Inhibitor (WRNi) GSK4418959 Alone or in Combination With Other Anti-cancer Agents in Adult Participants With Mismatch Repair-deficient (dMMR) or Microsatellite Instability-High (MSI-H) Solid Tumors (SYLVER)
Brief Title: A Study to Investigate the Safety, Pharmacokinetics, and Preliminary Effectiveness of GSK4418959 Alone or in Combination With Other Anti-cancer Agents in Participants With Solid Tumors
Acronym: SYLVER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 221971; 2024-519721-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Colorectal; Solid Tumor; Colon Cancer; Rectal Cancer; Endometrial Cancer
Keywords: GSK4418959; DNA Helicase Werner Inhibitor (WRNi); PD-1 inhibitor; Solid tumors; Colon cancer; Rectal cancer; Colorectal cancer; Endometrial cancer; Mismatch repair deficient; dMMR; microsatellite instability high; MSI-H
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Endometrial Neoplasms; Turcot syndrome | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: Dose escalation of GSK4418959 monotherapy (Experimental): Participants will receive GSK4418959 as monotherapy.
  Interventions: Drug: GSK4418959
- Part 2: Dose expansion of GSK4418959 monotherapy (Experimental): Participants will receive GSK4418959 as monotherapy.
  Interventions: Drug: GSK4418959
- Part 3: Dose escalation of GSK4418959 plus PD-1 inhibitor (Experimental): Participants will receive GSK4418959 plus PD-1 inhibitor.
  Interventions: Drug: GSK4418959; Biological: PD-1 inhibitor

INTERVENTIONS:
Drug: GSK4418959 — GSK4418959 will be administered.
Biological: PD-1 inhibitor — PD-1 inhibitor will be administered.
  Arms: Part 3: Dose escalation of GSK4418959 plus PD-1 inhibitor

SUMMARY:
Solid tumours are abnormal lumps of tissue that can occur in different parts of the body. The tumours involved in this study have specific genetic characteristics that can make them more aggressive and challenging to treat. The study will test whether GSK4418959 alone or in combination with a PD-1 inhibitor agent can decrease tumor size, is safe, well-tolerated, and how amounts of the study drug decrease in the body over time.

ELIGIBILITY:
Inclusion Criteria:

Parts 1, 2, and 3 inclusion criteria:

* Has a histologically diagnosed advanced (unresectable, metastatic or recurrent) solid tumor
* Has a known dMMR/MSI-H status as determined by a certified local laboratory at the time of Pre-screening or has an unknown Mismatch repair (MMR)/ Microsatellite Instability (MSI) status at the time of Pre-screening and MMR/MSI status will be determined by central reference laboratory
* Provides an archival or fresh (preferred) formalin fixed, paraffin embedded (FFPE) sample
* Intends to receive GSK4418959 (alone or in combination with PD-1 inhibitor, as determined between Investigator and sponsor) as next line of treatment
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Is expected to have a minimum of 3 months life expectancy
* Has adequate organ function, as defined in the protocol

Parts 1 and 3 inclusion criteria:

• Has histologically diagnosed advanced (unresectable, metastatic or recurrent) solid tumor and has exhausted all standard of care treatment options

Part 2 inclusion criteria:

* Has histologically diagnosed advanced (unresectable, metastatic or recurrent) Colorectal cancer (CRC) or Endometrial cancer (EC)
* Has received at least 1 but no more than 3 lines of systemic anticancer therapy for their advanced (unresectable, metastatic or recurrent) disease including at least one line of Immune checkpoint inhibitors (ICI) therapy
* Has measurable disease (i.e., at least 1 target lesion) during the Screening period per RECIST 1.1, as determined by the investigator

Exclusion Criteria:

Parts 1, 2, and 3 exclusion criteria:

* Has not recovered (i.e., to Grade ≤1 or to baseline) from prior anticancer therapy-induced AEs
* Has received prior treatment with a WRN inhibitor
* Is unable to swallow and retain orally administered study treatment
* Has symptomatic uncontrolled brain or leptomeningeal metastases
* Has a known additional malignancy that progressed or required active treatment within the last 2 years because reoccurrence of another malignancy would confound interpretation by RECIST 1.1 criteria. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cancer that is considered to be low risk for progression by the investigator
* Has any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs
* Has severe liver fibrosis
* Has cirrhosis or current unstable liver or biliary disease
* Has known hypersensitivity to any of the study interventions or any of their excipients
* Has known WRN syndrome
* Has an active autoimmune disease that has required systemic treatment in the past 2 years

Part 3 exclusion criteria:

* Has experienced any of the following with prior immunotherapy: any immune mediated adverse events (imAE) of Grade ≥3, immune-related severe neurologic events of any grade, exfoliative dermatitis of any grade (Stevens-Johnson Syndrome, toxic epidermal necrolysis, or Drug rash with eosinophilia and systemic signs syndrome [DRESS] syndrome), or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary
* Has any history of interstitial lung disease or pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with dose limiting toxicities (DLTs) during DLT observation period | Up to 21 days
Part 3: Number of participants with dose limiting toxicities (DLTs) during DLT observation period | Up to 21 days
Part 1: Number of participants with treatment emergent adverse events (TEAEs) during DLT observation period | Up to 21 days
Part 3: Number of participants with treatment emergent adverse events (TEAEs) during DLT observation period | Up to 21 days
Part 1: Number of participants with dosage interruptions, dose reductions, and drug discontinuations for TEAEs during DLT observation period | Up to 21 days
Part 3: Number of participants with dosage interruptions, dose reductions, and drug discontinuations for TEAEs during DLT observation period | Up to 21 days
Part 2: Objective Response Rate (ORR) | Up to approximately 26 months
  ORR is defined as percentage of participants with confirmed complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) by investigator assessment.

SECONDARY OUTCOMES:
Part 1: Area under the concentration-time curve (AUC) for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 1: Maximum concentration (Cmax) for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 1: Time to maximum concentration (Tmax) for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 3: AUC for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 3: Cmax for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 3: Tmax for GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)
Part 1: Number of participants with TEAEs | Up to approximately 42 months
Part 2: Number of participants with TEAEs | Up to approximately 42 months
Part 3: Number of participants with TEAEs | Up to approximately 42 months
Part 1: Number of participants with dosage interruptions, dose reductions, and drug discontinuations for TEAEs | Up to approximately 42 months
Part 2: Number of participants with dosage interruptions, dose reductions, and drug discontinuations for TEAEs | Up to approximately 42 months
Part 3: Number of participants with dosage interruptions, dose reductions, and drug discontinuations for TEAEs | Up to approximately 42 months
Part 1: Number of participants with clinical laboratory abnormalities | Up to approximately 42 months
Part 2: Number of participants with clinical laboratory abnormalities | Up to approximately 42 months
Part 3: Number of participants with clinical laboratory abnormalities | Up to approximately 42 months
Part 2: Progression-free Survival (PFS) | Up to approximately 42 months
  PFS is defined as time from first dose to progressive disease (as assessed per RECIST 1.1 by Investigator assessment) or death from any cause, whichever is earlier.
Part 2: Duration of Response (DoR) | Up to approximately 42 months
  DoR is defined as time from first documented PR or CR to progressive disease (as assessed per RECIST 1.1 by investigator assessment) or death from any cause, whichever is earlier for participants who have achieved a confirmed CR or PR.
Part 2: Plasma concentration of GSK4418959 | From first day of dosing for the duration of treatment until end of interventional phase (EOI) (up to approximately 42 months)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
- GSK Investigational Site, Melbourne, Victoria, Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Amsterdam, Netherlands
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/